CLINICAL TRIAL: NCT04462029
Title: A Randomized, Open-label, Single-dose, Crossover Study to Evaluate the Pharmacokinetics and Safety/Tolerability of BR4002 Comparing to BR4002-1 in Healthy Volunteers
Brief Title: A Study to Compare the Pharmacokinetics of BR4002 and BR4002-1 in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-DPZ-CT-102
Record Dates: First submitted 2020-07-01; First posted 2020-07-08 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Dementia Alzheimers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- sequence 1 (Other): A total of 18 subjects will be randomized into 6 sequence groups. The investigational products (IPs) will be administered according to the treatment groups (R, T1, and T2) assigned to each sequence group in Period 1, Period 2, and Period 3. In between each period, there will be a washout period (28 days) long enough for the administered IP to be metabolized and eliminated.
  * R(Reference): BR4002-1 (oral intake) 5mg single-dose
  * T1(Test1): BR4002 (patch) 5mg single-dose (using the applicator)
  * T2(Test2): BR4002 (patch) 5mg single-dose (not using the applicator)
  sequence 1: R - T1 - T2
  Interventions: Drug: BR4002; Drug: BR4002-1
- sequence 2 (Other): A total of 18 subjects will be randomized into 6 sequence groups. The investigational products (IPs) will be administered according to the treatment groups (R, T1, and T2) assigned to each sequence group in Period 1, Period 2, and Period 3. In between each period, there will be a washout period (28 days) long enough for the administered IP to be metabolized and eliminated.
  * R(Reference): BR4002-1 (oral intake) 5mg single-dose
  * T1(Test1): BR4002 (patch) 5mg single-dose (using the applicator)
  * T2(Test2): BR4002 (patch) 5mg single-dose (not using the applicator)
  sequence 2: R - T2 - T1
  Interventions: Drug: BR4002; Drug: BR4002-1
- sequence 3 (Other): A total of 18 subjects will be randomized into 6 sequence groups. The investigational products (IPs) will be administered according to the treatment groups (R, T1, and T2) assigned to each sequence group in Period 1, Period 2, and Period 3. In between each period, there will be a washout period (28 days) long enough for the administered IP to be metabolized and eliminated.
  * R(Reference): BR4002-1 (oral intake) 5mg single-dose
  * T1(Test1): BR4002 (patch) 5mg single-dose (using the applicator)
  * T2(Test2): BR4002 (patch) 5mg single-dose (not using the applicator)
  sequence 3: T1 - R - T2
  Interventions: Drug: BR4002; Drug: BR4002-1
- sequence 4 (Other): A total of 18 subjects will be randomized into 6 sequence groups. The investigational products (IPs) will be administered according to the treatment groups (R, T1, and T2) assigned to each sequence group in Period 1, Period 2, and Period 3. In between each period, there will be a washout period (28 days) long enough for the administered IP to be metabolized and eliminated.
  * R(Reference): BR4002-1 (oral intake) 5mg single-dose
  * T1(Test1): BR4002 (patch) 5mg single-dose (using the applicator)
  * T2(Test2): BR4002 (patch) 5mg single-dose (not using the applicator)
  sequence 4: T1 - T2 - R
  Interventions: Drug: BR4002; Drug: BR4002-1
- sequence 5 (Other): A total of 18 subjects will be randomized into 6 sequence groups. The investigational products (IPs) will be administered according to the treatment groups (R, T1, and T2) assigned to each sequence group in Period 1, Period 2, and Period 3. In between each period, there will be a washout period (28 days) long enough for the administered IP to be metabolized and eliminated.
  * R(Reference): BR4002-1 (oral intake) 5mg single-dose
  * T1(Test1): BR4002 (patch) 5mg single-dose (using the applicator)
  * T2(Test2): BR4002 (patch) 5mg single-dose (not using the applicator)
  sequence 5: T2 - R - T1
  Interventions: Drug: BR4002; Drug: BR4002-1
- sequence 6 (Other): A total of 18 subjects will be randomized into 6 sequence groups. The investigational products (IPs) will be administered according to the treatment groups (R, T1, and T2) assigned to each sequence group in Period 1, Period 2, and Period 3. In between each period, there will be a washout period (28 days) long enough for the administered IP to be metabolized and eliminated.
  * R(Reference): BR4002-1 (oral intake) 5mg single-dose
  * T1(Test1): BR4002 (patch) 5mg single-dose (using the applicator)
  * T2(Test2): BR4002 (patch) 5mg single-dose (not using the applicator)
  sequence 6: T2 - T1 - R
  Interventions: Drug: BR4002; Drug: BR4002-1

INTERVENTIONS:
Drug: BR4002 — * Administration to the T1 group: 5 mg of BR4002 (patch) will be attached using an applicator for 24 hours
  * Administration to the T2 group: 5 mg of BR4002 (patch) will be attached without using an applicator for 24 hours
Drug: BR4002-1 — Administration to the R group: 5 mg of BR4002-1 (oral formulation) will be administered with 150 mL of water

SUMMARY:
This study is designed as a randomized, open-label, single-dose, 6x3 crossover study.

DETAILED DESCRIPTION:
A total of 18 subjects will be randomized into 6 sequence groups. The investigational products will be administered according to the treatment groups (R, T1, and T2) assigned to each sequence group in Period 1, Period 2, and Period 3. In between each period, there will be a washout period (28 days) long enough for the administered IP to be metabolized and eliminated.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged ≥ 19 and ≤ 55 years at screening
2. Body weight of ≥ 50 kg with calculated body mass index (BMI) of ≥ 18.0 to ≤ 29.0 kg/m2
3. Determined eligible based on the results of physical examination and investigator questioning conducted according to this protocol. That is, absence of congenital or chronic disease, and absence of pathological symptoms or findings based on medical examination in the last 3 years.
4. Determined eligible based on the results of the laboratory tests and electrocardiogram (ECG) conducted according to this protocol
5. Voluntarily decided to participate in the study and provided written consent to follow precautions after receiving a detailed explanation on this study and fully understanding the information

Exclusion Criteria:

1. Hypersensitivity to, or history of clinically significant hypersensitivity to donepezil hydrochloride, piperidine derivatives or any ingredients of piperidine derivatives, or other drugs (aspirin, antibiotics, etc.)
2. Hereditary disorders including galactose intolerance, Lapp lactase deficiency, and glucose-galactose malabsorption
3. History of heart disease such as sinus node syndrome, intra-atrial conduction disturbance or atrioventricular junctional conduction disturbance
4. Ongoing administration of non-steroidal anti-inflammatory drugs or history of peptic ulcer
5. History of asthma or obstructive pulmonary disease
6. Extrapyramidal disorder
7. Psychotic disorders or drug addiction
8. Presence or prior history of a gastrointestinal disorder or prior history of gastrointestinal surgery or skin graft that may affect the absorption of the IP
9. Presence or prior history of clinically significant cardiovascular, respiratory, hepatic, renal, neurological, endocrine, hematological and oncological, psychotic, or urinary disease
10. Clinically significant hypotension (systolic blood pressure < 90 mmHg) or hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 95 mmHg) at screening
11. Any of the following results from screening tests:

    * AST or ALT > 2 times the upper limit of normal
    * Total bilirubin > 2.0 mg/dL
    * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2
12. QTc > 450 ms or any clinically significant abnormal finding from an ECG result at screening
13. Continuous alcohol intake or inability to stop drinking during the study period
14. Continuous smoking or inability to stop smoking throughout the hospitalization during the study period
15. Participated in another clinical study or bioequivalence study within 6 months prior to the first administration of the IP
16. Donated whole blood within 60 days or blood components within 30 days, or received blood transfusion within 30 days prior to the first administration of the IP
17. Used any prescription drugs or herbal medicines within 14 days, or any over-the-counter (OTC) drugs within 7 days prior to the first administration of the IP
18. Used drugs inducing and inhibiting drug-metabolizing enzymes, such as barbitals, within 1 month prior to initiation of the study
19. Have been on a diet (especially grapefruit juice or its product) which may affect absorption, distribution, metabolism, and excretion of the drug within 7 days prior to the first administration of the IP
20. Do not agree to exclude the possibility of pregnancy by using medically acceptable methods of contraception from the first day of administration of the IP up to 7 days after the last day of administration of the IP
21. Unwillingness or inability to comply with the diet and lifestyle guidelines required for the study
22. Clinically significant abnormal laboratory results or considered ineligible for study participation by the investigator for any other reason
23. Women who are pregnant, have a positive serum/urine hCG test, or are breastfeeding

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables -Area Under the concentration-time Curve from time 0 to t after single dosing(AUCt) of BR4002 and BR4002-1 | 0~240 hours after medication
  PK data of subjects who complete all of the scheduled blood collections without any major protocol deviations considered to affect the PK results after administration of the IP and have quantifiable drug concentrations for PK assessment will be analyzed.
Pharmacokinetic variables - maximum observed plasma concentration(Cmax) of BR4002 and BR4002-1 | 0~240 hours after medication
  PK data of subjects who complete all of the scheduled blood collections without any major protocol deviations considered to affect the PK results after administration of the IP and have quantifiable drug concentrations for PK assessment will be analyzed.

SECONDARY OUTCOMES:
Pharmacokinetic variables - Area Under the concentration-time Curve from time 0 to infinite after single dosing(AUCinf) of BR4002 and BR4002-1 | 0~240 hours after medication
  PK data of subjects who complete all of the scheduled blood collections without any major protocol deviations considered to affect the PK results after administration of the IP and have quantifiable drug concentrations for PK assessment will be analyzed.
Pharmacokinetic variables - Time of occurrence of Cmax(Tmax) of BR4002 and BR4002-1 | 0~240 hours after medication
  PK data of subjects who complete all of the scheduled blood collections without any major protocol deviations considered to affect the PK results after administration of the IP and have quantifiable drug concentrations for PK assessment will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Heon Cho, Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea